CLINICAL TRIAL: NCT02632305
Title: A Multicentre, Open-label Phase II Study of Nab-paclitaxel in Combination With Gemcitabine + Cisplatin as First Line Treatment in Patients With Unresectable Biliary Tract Cancer
Brief Title: A Study to See the Effects That a New Combination of the Three Drugs, Nab-paclitaxel, Gemcitabine, and Cisplatin Has on Biliary Tract Cancer
Acronym: AX-CSARC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AX-CSARC-PI-0001
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Biliary Tract Cancer
Keywords: unresectable biliary tract cancer; nab-paclitaxel; cisplatin; gemcitabine
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Eligible patients will receive nab-paclitaxel in combination with gemcitabine + cisplatin at the recommended phase II dose based on the phase I study completed in metastatic pancreas cancer patients.
  The doses of study drugs will be as follows:
  * nab-Paclitaxel 100 mg/m2 day 1 and 8 every 21 days
  * Cisplatin 25 mg/m2 day 1 and 8 every 21 days
  * Gemcitabine 800 mg/m2 day 1 and 8 every 21 days
  Nab-paclitaxel will be administered first followed by cisplatin and then gemcitabine on day 1 and 8 of each treatment cycle. Cycles will be 3 weeks in length (21 days).
  Interventions: Drug: nab-paclitaxel in combination with gemcitabine + cisplatin

INTERVENTIONS:
Drug: nab-paclitaxel in combination with gemcitabine + cisplatin — Patients with unresectable BTC will be treated with the triple combination of nab-paclitaxel in combination with gemcitabine + cisplatin

SUMMARY:
You are being asked to take part in this study because you have a biliary cancer that is incurable and has spread to other organs. Chemotherapy is often used to help shrink the cancer temporarily and may improve survival. In Canada, the combination of gemcitabine and cisplatin is the chemotherapy combination used to treat biliary cancer that has spread. There is no other known treatment for biliary cancer that has spread to other organs. It is hoped that this new combination of drugs (nab-paclitaxel, gemcitabine, and cisplatin) will improve the tumor shrinkage rate.

This study is being done because we do not know whether 2 or 3 chemotherapy drugs is better to treat biliary cancers.

We hope to learn whether giving nab-paclitaxel, gemcitabine, and cisplatin together in patients with biliary cancer can increase tumor shrinkage without too many side effects.

The purpose of this study is to find out what effects (good and bad) nab-paclitaxel, gemcitabine, and cisplatin has on you and your biliary cancer.

DETAILED DESCRIPTION:
There is increasing evidence that there is a large degree of pathologic homology between the pancreas and biliary tract. Indeed, the biliary tract has been referred to as "an incomplete pancreas" and embryologically the two originate from the same structure. It is thus plausible that oncogenesis in the pancreas and biliary tract are related and that pancreas and biliary cancers have reciprocal effective treatment strategies.

To date, the only chemotherapeutic agents effective in advanced biliary tract tumors is the combination of gemcitabine and cisplatin. Known and approved therapies for advanced pancreas cancer include single agent gemcitabine, the four drug combination of FOLFIRINOX (5-fluorouracil, leucovorin, oxaliplatin, and irinotecan), the questionable limited benefit of inhibiting the epidermal growth factor receptor pathway, and most recently the combination of gemcitabine and nab-paclitaxel.

Based on promising results in pancreas cancer, investigators hypothesize nab-paclitaxel in combination with gemcitabine + cisplatin will be an effective cytotoxic combination in BTC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented locally advanced or metastatic BTC (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer, or ampullary carcinoma) not previously treated with palliative systemic therapy or radiation
2. Unresectable disease based on the presence of clinically and/or radiologically documented measurable disease based on RECIST 1.1. Patients must have measurable disease; evaluable only disease will not be permitted.
3. ECOG performance status of 0 - 1.
4. Age ≥ 18 years.
5. Life expectancy of at least 3 months based on discretion of treating oncologist.
6. Adequate hematologic function defined by the following laboratory parameters:

   * Hemoglobin ≥ 9 g/dL
   * Platelet count ≥ 100 x 109/L
   * Absolute granulocyte count ≥ 1.5 x 109/L
7. Adequate hepatic and renal function defined by the following laboratory parameters:

   * AST and ALT and alkaline phosphatase ≤ 2.5 X upper limit of institutional normal (≤ 5 if liver metastases)
   * bilirubin ≤ 1.5 X upper limit of institutional normal
   * serum creatinine ≤ upper limit of institutional normal OR calculated creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault formula
8. Patients may have received prior surgery if this surgery was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
9. Prothrombin time- international normalized ratio (PT-INR) and partial thromboplastin time (PTT) must be within +/- 15% normal range.
10. Patients who have treated brain metastasis (via local radiation standards or surgical resection or local ablative techniques) and who are either off steroids or on a stable dose of steroids for at least one month (30 days), AND who are off anticonvulsants, AND have radiological documented stability of lesions for at least 3 months may be eligible. Each case should be discussed with the study Chair.
11. Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.
12. Female subjects of childbearing potential, defined as a sexually mature woman who 1) has not undergone hysterectomy or bilateral oophorectomy OR 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time during the preceding 24 consecutive months) must:

    * either commit to true abstinence or agree to the use of a 2 physician-approved contraceptive methods (oral, injectable, or implantable hormonal contraceptive with spermicide; or vasectomized partner) while on clinical trial and for at least 3 months following the last does of study medication; and
    * has a negative serum pregnancy test (β-hCG) result at screening. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 6 months following study medication discontinuation, even if he has undergone a success vasectomy.

Exclusion Criteria:

1. Patients who have received prior palliative chemotherapy for their advanced BTC.
2. Prior curative or palliative radiation treatment to the pelvis or radiation therapy to ≥ 25% of bone marrow stores.
3. History of bowel obstruction due to peritoneal metastases or clinically documented ascites requiring paracenteses.
4. Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or uterus or non-melanoma skin cancer or in-situ carcinoma of the prostate (Gleason score ≤ 7, with all treatment being completed 6 months prior to enrollment, unless at least 5 years have elapsed since last treatment and the patient is considered cured).
5. Active bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
6. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications.
7. Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, cerebrovascular diseases, uncontrolled hypertension, uncontrolled diabetes, uncontrolled psychiatric disorder, serious infection, active peptic ulcer disease, or other medical condition that may be aggravated by treatment.
8. Pre-existing neuropathy ≥ grade 1 from any cause.
9. Patients with unstable metastasis to the central nervous system (CNS). A CT scan or MRI is NOT required to rule out brain metastases unless there is clinical suspicion of CNS involvement.
10. Pregnant or lactating women; women of child bearing potential must have a negative serum pregnancy test within 7 days of trial registration. Women or men of child bearing potential must use effective contraception (defined by the treating physician) which must be documented in study CRFs.
11. History of allergic reaction to planned study medications.
12. Patient has a ≥ 20% decrease in serum albumin level between baseline visit, if available, and within 72 hours prior to first study treatment dose.
13. Patient is on coumadin.
14. History of interstitial lung disease.
15. History of connective tissue disorders (e.g. lupus, scleroderma, polyarteritis nodosa).
16. Enrollment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.
17. Any significant medical condition, laboratory abnormality, or psychiatric illness, that would prevent the subject from participating in the study, places the subject at unacceptable risk if he/she were to participate in the study, or any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rates | 1 year
  defined as the sum of complete response rates and partial response rates, of nab-paclitaxel in combination with gemcitabine + cisplatin in first line treatment of unresectable biliary tract cancer (BTC).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Spratlin, MD FRCPC, Principal Investigator — Alberta Health services
Locations (2):
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No